CLINICAL TRIAL: NCT00268333
Title: Phase II Study of Recurrent Ganglionic Colorectal Cancer Not Accessible By Surgery Treated Using Chemotherapy With Simplified FOLFOX7 Followed By Radiotherapy Combined With 5FU and Oxaliplatin
Brief Title: Combination Chemotherapy and Radiation Therapy in Treating Patients With Recurrent Metastatic Colorectal Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GERCOR - Multidisciplinary Oncology Cooperative Group (Other)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Non-Randomized | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000453784; GERCOR-C04-1; EU-20568; SANOFI-GERCOR-C04-1
Record Dates: First submitted 2005-12-20; First posted 2005-12-22 (Estimated); Last update posted 2009-02-09 (Estimated); Status verified 2007-05

CONDITIONS: Colorectal Cancer
Keywords: adenocarcinoma of the colon; adenocarcinoma of the rectum; stage IV colon cancer; stage III colon cancer; stage III rectal cancer; stage IV rectal cancer
MeSH Terms: conditions — Colorectal Neoplasms; Colonic Neoplasms; Rectal Neoplasms | interventions — Fluorouracil; Leucovorin; Oxaliplatin; Neoadjuvant Therapy

INTERVENTIONS:
Drug: fluorouracil
Drug: leucovorin calcium
Drug: oxaliplatin
Procedure: neoadjuvant therapy

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as oxaliplatin, fluorouracil, and leucovorin, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Radiation therapy uses high-energy x-rays to kill tumor cells. Giving more than one drug (combination chemotherapy) together with radiation therapy may kill more tumor cells.

PURPOSE: This phase II trial is studying how well giving combination chemotherapy together with radiation therapy works in treating patients with recurrent metastatic colorectal cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the response rate in patients with recurrent metastatic colorectal cancer treated with neoadjuvant oxaliplatin, fluorouracil, and leucovorin calcium followed by radiotherapy and concurrent fluorouracil and oxaliplatin.

Secondary

* Determine the overall survival and disease-free survival of patients treated with this regimen.
* Determine the primary site of recurrence and time to recurrence in patients treated with this regimen.
* Determine quality of life of patients treated with this regimen.

OUTLINE: This is a nonrandomized, open-label, multicenter study.

* Neoadjuvant chemotherapy: Patients receive oxaliplatin IV over 2 hours and leucovorin calcium IV over 2 hours on day 1. Patients also receive fluorouracil IV continuously over 46 hours beginning day 1. Treatment repeats every 14 days for 4 courses in the absence of disease progression or unacceptable toxicity. Two to 5 weeks later, patients with stable or responding disease proceed to chemoradiotherapy.
* Chemoradiotherapy: Patients receive fluorouracil IV continuously 5 days a week for 5 weeks and oxaliplatin IV over 1 hour on days 1, 8, 15, 22, and 29. Patients also undergo radiotherapy 5 days a week for 5 weeks beginning on day 1.

Quality of life is assessed at baseline, 1 week after the completion of neoadjuvant chemotherapy, on days 15, 30, and 42 of chemoradiotherapy, and at 1 and 2 months after the completion of study treatment.

After completion of study treatment, patients are followed periodically.

PROJECTED ACCRUAL: A total of 39 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed adenocarcinoma of the colon or rectum

  * Metastatic disease isolated to the following lymph nodes:

    * Aortic
    * Interaortic
    * Celiomesenteric
    * Retroperitoneal, including the following sites:

      * Peri-uretal
      * Liver
      * Iliac
      * Clavicle
      * Mediastinum
      * Inguinal
      * Cervical
* Incompletely resected disease
* Recurrent disease, defined by 1 of the following criteria:

  * Progression occurred within 6 months after prior oxaliplatin or after the patient received no prior oxaliplatin
  * Progressive disease after cisplatin or fluorouracil
* Must be able to be encompassed in radiation field

PATIENT CHARACTERISTICS:

* ECOG performance status (PS) 0-2 or Karnofsky PS 60-100%
* Life expectancy more than 12 weeks
* Absolute neutrophil count ≥ 1,500/mm^3
* Platelet count ≥ 100,000 /mm^3
* Alkaline phosphatase ≤ 5 times normal
* Bilirubin ≤ 2 times normal
* Creatinine < 2 times normal or creatinine clearance ≥ 40 mL/min
* No peripheral neuropathy > grade 1
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No weight loss > 15% since diagnosis of recurrent disease
* No uncontrolled heart disease
* No angina
* No symptomatic disease of the inferior artery
* No psychological, familial, sociological, or geographical condition that would preclude study treatment or compliance

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* No prior chemotherapy or radiotherapy
* No concurrent corticosteroids

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Estimated)
Dates: Start 2005-08; Primary Completion 2006-01 (Actual)

PRIMARY OUTCOMES:
Response rate

SECONDARY OUTCOMES:
Overall survival
Disease-free survival
Primary site of recurrence
Time to recurrence
Quality of life

CONTACTS AND LOCATIONS:
Overall Officials: Laurent Mineur, MD, Study Chair — Institut Sainte Catherine
Locations (9):
- France (9):
  - Institut Sainte Catherine, Avignon
  - Centre Hospitalier Regional de Besancon - Hopital Jean Minjoz, Besançon
  - Hopital Drevon, Dijon
  - Hopital Robert Boulin, Libourne
  - Polyclinique des Quatre Pavillons, Lormont
  - Hopital Europeen Georges Pompidou, Paris
  - Hopital Tenon, Paris
  - Polyclinique De Courlancy, Reims
  - C.H. Senlis, Senlis